CLINICAL TRIAL: NCT07083063
Title: Precise Endoscopic Application of Nitroglycerin in Preventing Post-ERCP Pancreatitis: A Randomized Controlled Trial
Brief Title: Precise Endoscopic Application of Nitroglycerin in Preventing Post-ERCP Pancreatitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Hsueh-Chien Chiang, Medical Doctor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-BR-114-025
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-07

CONDITIONS: Pancreatitis
Keywords: post-ERCP pancreatitis; nitroglycerin
MeSH Terms: conditions — Pancreatitis | interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Intervention Model Description: All patients without chronic kidney disease (serum creatine > 1.5 mg/dL) will receive rectal diclofenac 100 mg before the procedure. During the biliary cannulation, if twice or more times of pancreatic duct cannulation, a pancreatic plastic stent will be placed. Lactate ringer hydration with standard dose (1.5 kg/cc/hr) will be provided to patients with pancreatic duct cannulation for 8 hours. After the EST and stone extraction, we will randomly assign the patients to either a control or an intervention group. After EST, if immediate bleeding occurs, investigators will apply standard endoscopic therapy by either local injection of diluted epinephrine or heater probe coagulation. Before the end of the exam, diluted 1mg nitroglycerin in normal saline (1mg/10cc) will be delivered to the major papilla in the intervention group. Normal saline 10cc will be delivered to the major papilla in the standard group.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): diluted 1mg nitroglycerin in normal saline (1mg/10cc) will be delivered to the major papilla in the intervention group.
  Interventions: Drug: Nitroglycerin (NTG)
- Standard Group (Placebo Comparator): 10cc normal saline will be delivered to the major papilla in the standard group.
  Interventions: Drug: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Nitroglycerin (NTG) — All patients without chronic kidney disease (serum creatine > 1.5 mg/dL) will receive rectal diclofenac 100 mg before the procedure. During the biliary cannulation, if twice or more times of pancreatic duct cannulation, a pancreatic plastic stent will be placed. Lactate ringer hydration will be provided to patients with pancreatic duct cannulation for 24 hours. After the EST and stone extraction, we will randomly assign the patients to either a control or an intervention group. After EST, if immediate bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine or heater probe coagulation. Before the end of the exam, diluted 1mg nitroglycerin in normal saline (1mg/10cc) will be delivered to the major papilla in the intervention group, and 10cc normal saline will be delivered to the major papilla in the standard group.
  Arms: Intervention Group
Drug: Normal Saline (0.9% NaCl) — All patients without chronic kidney disease (serum creatine > 1.5 mg/dL) will receive rectal diclofenac 100 mg before the procedure. During the biliary cannulation, if twice or more times of pancreatic duct cannulation, a pancreatic plastic stent will be placed. Lactate ringer hydration will be provided to patients with pancreatic duct cannulation for 24 hours. After the EST and stone extraction, we will randomly assign the patients to either a control or an intervention group. After EST, if immediate bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine or heater probe coagulation. Before the end of the exam, diluted 1mg nitroglycerin in normal saline (1mg/10cc) will be delivered to the major papilla in the intervention group.
  Arms: Standard Group

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a technically demanding procedure combining endoscopy and fluoroscopy to diagnose and treat pancreaticobiliary disorders such as bile duct stones, strictures, and cholangitis. Despite its therapeutic value, ERCP carries a relatively high complication risk of about 10%, with severe complications occurring in roughly 24% of those affected and mortality rates between 0.2% and 0.7%. The most common and significant complication is post-ERCP pancreatitis (PEP), occurring in 2% to 10% of average patients and up to 40% or higher in high-risk groups. PEP ranges from mild, self-limiting inflammation to severe, life-threatening conditions including pancreatic necrosis and multi-organ failure.

PEP arises from mechanical trauma, hydrostatic injury, chemical irritation, or infection during ERCP that activates inflammatory pathways within the pancreas. Key patient-related risk factors include young age, female sex, prior pancreatitis, and sphincter of Oddi dysfunction; procedural factors include difficult biliary cannulation, pancreatic duct manipulation, and precut sphincterotomy.

Preventive strategies focus on minimizing mechanical injury and pharmacologic prophylaxis. Rectal NSAIDs (indomethacin, diclofenac) administered immediately before ERCP are well-supported for reducing PEP risk. Periprocedural aggressive intravenous hydration and prophylactic pancreatic duct stenting in high-risk cases also lower PEP incidence.

Nitroglycerin, a smooth muscle relaxant acting via nitric oxide-mediated sphincter relaxation, has shown promise in PEP prevention, especially in patients contraindicated for NSAIDs. Clinical trials indicate that transdermal or sublingual nitroglycerin reduces PEP rates, and combined use with NSAIDs may enhance protection. However, current guidelines do not routinely recommend nitroglycerin due to limited consensus on its efficacy.

Topical nitroglycerin, known to relax smooth muscles locally and used in anorectal conditions, might reduce sphincter of Oddi pressure without systemic side effects. This suggests potential benefit in lowering PEP incidence or severity when applied topically during ERCP, pending further investigation. This study aimed to investigate whether topical delivery of nitroglycerin can reduce the incidence rate of PEP or the severity of pancreatitis.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is a complex procedure that combines endoscopy and fluoroscopy for the diagnosis and treatment of pancreaticobiliary ductal disorders, such as choledocholithiasis (bile duct stones), biliary strictures, and cholangitis (bile duct inflammation). Although ERCP is vital for both diagnosis and treatment, it carries a higher risk of complications than do other endoscopic procedures. Common complications include post-ERCP pancreatitis (PEP), bleeding, perforation, and biliary tract infections. The overall incidence rate of ERCP-associated complications is approximately 10%, with severe complications occurring in about 24% of patients who experience any complications. The rate of ERCP-associated mortality ranges from 0.2% to 0.7%. Despite technological advancements and enhanced safety protocols, the rate of ERCP-associated complications remains high.

Among all complications, post-ERCP pancreatitis presents a major challenge for clinicians and endoscopists. PEP increased hospitalization interval and mortality. While most cases of PEP are mild and resolve with conservative treatment, it can be dangerous in severe cases, such as pancreatic necrosis, multi-organ failure, and peripancreatic fluid collections. These complications are rare but can be fatal. The incidence rate of PEP varies depending on the patient population and risk factors. Generally, the overall incidence of PEP is reported to be between 2% and 10% in unselected patient samples. However, in high-risk patients, this rate can increase significantly, ranging from 8% to 40% or even higher. High-risk patients for post-ERCP pancreatitis include several groups based on both patient-related and procedure-related factors. Patient-related risk factors include female gender, younger patients under 50 years old, history of pancreatitis, and sphincter of Oddi dysfunction. Procedure-related risk factors include difficult biliary cannulation, precut papillotomy, and pancreatic duct cannulation.

Preventing PEP involves several strategies that can be implemented before, during, and after the procedure. Rectal nonsteroidal anti-inflammatory drugs (NSAIDs), such as indomethacin or diclofenac, should be administered immediately before ERCP to reduce the risk of PEP. High-volume intravenous fluids should be administered peri-procedurally to help prevent PEP. For high-risk patients with sphincter of Oddi dysfunction, difficult cannulation, or when the pancreatic duct is accessed repeatedly, prophylactic pancreatic stent placement during the procedure can reduce the risk of PEP.

Despite these preventing strategies, some patients still suffer from PEP. Additionally, patients with chronic kidney disease are contraindicated from NSAIDs. Instead, nitroglycerin has been shown to have a significant benefit in preventing PEP. Nitroglycerin plays a crucial role in managing angina pectoris for decades. Nitroglycerin affects smooth muscle primarily through its conversion to nitric oxide, which acts as a potent vasodilator. Nitric oxide activates the enzyme guanylate cyclase, which converts guanosine triphosphate (GTP) into cyclic guanosine monophosphate (cGMP), leading to protein kinase-dependent phosphorylation and activation of downstream cascades that promote relaxation of smooth muscle cells. Pancreatic sphincter hypertension increases the risk of PEP. In this situation, nitroglycerin could lower the basal pressure in the sphincter of Oddi and depress the resistance of bile outflow, which may be potential in preventing PEP.

Previous clinical trial demonstrated that 15mg transdermal nitroglycerin patch protects against post-ERCP pancreatitis. Another clinical trial revealed that 5 mg sublingual nitroglycerin 5 minutes before ERCP could reduce pancreatitis and hyperamylasemia. The combination use of rectal indomethacin and 0.5 mg sublingual nitroglycerin can also prevent and relieve the severity of PEP after ERCP in patients with difficult cannulation. Systemic review and meta-analysis studies confirmed that patients who received nitroglycerin were 39 % less likely to develop pancreatitis, suggesting that nitroglycerin administered by the sublingual or transdermal route may be useful. However, current guideline doesn't suggest routine use of nitroglycerin due to inadequate evidence of benefits.

In order to enhance the smooth muscle relaxation without inducing systemic adverse events, topical administration of nitroglycerin can be a good solution. Topical nitroglycerin has shown benefits in reducing the anal tone for patients with Levator ani syndrome. Topical nitroglycerin also demonstrated effects in relieving pain for patients with anal fissure. Reducing sphincter spasm could also reduce post-hemorrhoidectomy pain. From above evidence, topical administration of nitroglycerin has shown local effect of smooth muscle relaxation, which may be beneficial in reducing the PEP rate or severity. This study aimed to investigate whether topical delivery of nitroglycerin can reduce the incidence rate of PEP or the severity of pancreatitis.

Study design and rationale Participants will be recruited from the volunteers with choledocholithiasis at National Cheng Kung University Hospital. Eligible participants include patients aged ≥ 18 years who accept ERCP and sphincterotomy for common bile duct (CBD) stone extraction. Patient consent forms will be given and explained to all patients before the ERCP. Exclusion criteria include patients with pancreatic cancer, shock status (systolic blood pressure < 90 mmHg or using inotropic agents), allergy to NTG, angle-closure glaucoma, severe anemia, and patients on PDE 5 inhibitors. After patient enrollment, investigators will randomize the patient into either the intervention group or control group by sealed envelope randomization method.

All patients without chronic kidney disease (serum creatine > 1.5 mg/dL) will receive rectal diclofenac 100 mg before the procedure. During the biliary cannulation, if twice or more times of pancreatic duct cannulation, a pancreatic plastic stent will be placed. Lactate ringer hydration will be provided to patients with pancreatic duct cannulation for 24 hours. After the EST and stone extraction, investigators will randomly assign the patients to either a control or an intervention group. After EST, if immediate bleeding occurs, investigators will apply standard endoscopic therapy by either local injection of diluted epinephrine or heater probe coagulation. Before the end of the exam, diluted 1mg nitroglycerin in normal saline (1mg/10cc) will be delivered to the major papilla in the intervention group.

Blood tests A blood sample is obtained as ward routine to measure creatinine, albumin, total bilirubin, hemoglobin, lipase, platelet, prothrombin time (PT), and activated partial thromboplastin time (APTT). All lab data are checked by the central laboratory of the National Cheng Kung University Hospital.

Outcome measures All patients will be monitored for 14 days after the ERCP. The primary endpoint is the incidence rate of post-ERCP pancreatitis, which is defined as epigastric pancreatic pain with elevated serum lipase over 200 U/L. The secondary endpoints include (1) the level of serum lipase the day after ERCP; (2) length of hospitalization; (3) all-cause mortality.

Statistical analysis According to previous literature, investigators set the event rate of PEP is 20 % and the delivery of nitroglycerin can reduce the PEP rate to 10%. Investigators need to enroll 199 patients at least in each group to reject the null hypothesis that the effects are equal between the two groups with the probabilities of power at 0.8 and type I error at 0.05. Assuming a drop rate of 10%, this study will enroll a total of 440 patients, including 220 patients in the intervention group and 220 patients in the control group, respectively. Data related to baseline characteristics and the endpoints are evaluated using the Student's test, Pearson's χ2 test or Fisher's exact test, and the Mann-Whitney U test. All tests are two-tailed and P-values < 0.05 indicated significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include patients aged ≥ 18 years who accept ERCP and sphincterotomy for common bile duct (CBD) stone extraction.

Exclusion Criteria:

* patients with pancreatic cancer
* shock status (systolic blood pressure < 90 mmHg or using inotropic agents)
* allergy to NTG
* angle-closure glaucoma
* severe anemia
* patients on PDE 5 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Post-ERCP pancreatitis | 7 days
  Incidence of Post-ERCP pancreatitis based on a widely recognised Cotton consensus, which is defined as a three-fold increase of serum lipase at ≥24 h and necessitating hospital admission or prolonged hospital stay.

SECONDARY OUTCOMES:
Occurence of moderate or severe PEP | 7 days
  The severity classification of PEP was also defined according to the Cotton criteria. The categories included: (1) mild: an extension of hospitalisation period of 2-3 days; (2) moderate: an extension of hospitalisation period of 4-10 days; (3) severe: an extension of at least 10 days, or haemorrhagic pancreatitis, phlegmon or pseudocyst, intervention (percutaneous drainage or surgery) or death.
Occurrence of post-ERCP bleeding | 14 days
  All patients were monitored for 14 days after EST, either during hospitalization or outpatient follow-up. For patients reporting hematemesis or presenting with tarry or bloody stool, diagnostic endoscopy was performed to identify the source of bleeding.
Occurrence of shock status | 1 day
  Hypotension with SBP < 90mmHg or in need of inotropic agents after the application of NTG.
Length of hospitalization | 14 days
  Length of hospitalization
Level of pancreatic serology | 8 hours
  Serum lipase and amylase will be obtained on the 8 hours after ERCP

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Other (Non U.s.), Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Jin J, Unasa H, Bahl P, Mauiliu-Wallis M, Svirskis D, Hill A. Can Targeting Sphincter Spasm Reduce Post-Haemorrhoidectomy Pain? A Systematic Review and Meta-Analysis. World J Surg. 2023 Feb;47(2):520-533. doi: 10.1007/s00268-022-06807-3. Epub 2022 Nov 10. PMID 36357803
- [Result] Hussain S, Ammar AS, Hameed AR, Aslam I, Afzal A. Comparison of outcome of botulinum toxin injection with and without glyceryl trinitrate in chronic anal fissure in terms of post operative pain and healing. J Pak Med Assoc. 2024 Jul;74(7):1245-1248. doi: 10.47391/JPMA.9726. PMID 39028048
- [Result] Khan SS, Martin S, Doh CY, Stein SL, Steinhagen E. Trends in Management of Anal Fissures. Am Surg. 2024 Mar;90(3):393-398. doi: 10.1177/00031348231200662. Epub 2023 Sep 2. PMID 37658717
- [Result] Canlikarakaya F, Ocakli S. Can Topical Glyceryl Trinitrate be Effective in the Treatment of Levator Ani Syndrome? Turk J Gastroenterol. 2025 Jan 13;36(5):328-327. doi: 10.5152/tjg.2025.24489. PMID 39840843
- [Result] Kubiliun NM, Adams MA, Akshintala VS, Conte ML, Cote GA, Cotton PB, Dumonceau JM, Elta GH, Fogel EL, Freeman ML, Lehman GA, Naveed M, Romagnuolo J, Scheiman JM, Sherman S, Singh VK, Elmunzer BJ; United States Cooperative for Outcomes Research in Endoscopy (USCORE). Evaluation of Pharmacologic Prevention of Pancreatitis After Endoscopic Retrograde Cholangiopancreatography: A Systematic Review. Clin Gastroenterol Hepatol. 2015 Jul;13(7):1231-9; quiz e70-1. doi: 10.1016/j.cgh.2014.11.038. Epub 2015 Jan 9. PMID 25579870
- [Result] Bai Y, Xu C, Yang X, Gao J, Zou DW, Li ZS. Glyceryl trinitrate for prevention of pancreatitis after endoscopic retrograde cholangiopancreatography: a meta-analysis of randomized, double-blind, placebo-controlled trials. Endoscopy. 2009 Aug;41(8):690-5. doi: 10.1055/s-0029-1214951. Epub 2009 Aug 10. PMID 19670137
- [Result] Wang Y, Xu B, Zhang W, Lin J, Li G, Qiu W, Wang Y, Sun D, Wang Y. Prophylactic effect of rectal indomethacin plus nitroglycerin administration for preventing pancreatitis after endoscopic retrograde cholangiopancreatography in female patients. Ann Palliat Med. 2020 Nov;9(6):4029-4037. doi: 10.21037/apm-20-1963. PMID 33302662
- [Result] Hao JY, Wu DF, Wang YZ, Gao YX, Lang HP, Zhou WZ. Prophylactic effect of glyceryl trinitrate on post-endoscopic retrograde cholangiopancreatography pancreatitis: a randomized placebo-controlled trial. World J Gastroenterol. 2009 Jan 21;15(3):366-8. doi: 10.3748/wjg.15.366. PMID 19140238
- [Result] Nojgaard C, Hornum M, Elkjaer M, Hjalmarsson C, Heyries L, Hauge T, Bakkevold K, Andersen PK, Matzen P; European Post-ERCP Pancreatitis Preventing Study Group. Does glyceryl nitrate prevent post-ERCP pancreatitis? A prospective, randomized, double-blind, placebo-controlled multicenter trial. Gastrointest Endosc. 2009 May;69(6):e31-7. doi: 10.1016/j.gie.2008.11.042. PMID 19410035
- [Result] Kaffes AJ, Bourke MJ, Ding S, Alrubaie A, Kwan V, Williams SJ. A prospective, randomized, placebo-controlled trial of transdermal glyceryl trinitrate in ERCP: effects on technical success and post-ERCP pancreatitis. Gastrointest Endosc. 2006 Sep;64(3):351-7. doi: 10.1016/j.gie.2005.11.060. Epub 2006 May 19. PMID 16923481
- [Result] Moreto M, Zaballa M, Casado I, Merino O, Rueda M, Ramirez K, Urcelay R, Baranda A. Transdermal glyceryl trinitrate for prevention of post-ERCP pancreatitis: A randomized double-blind trial. Gastrointest Endosc. 2003 Jan;57(1):1-7. doi: 10.1067/mge.2003.29. PMID 12518122
- [Result] Kochar B, Akshintala VS, Afghani E, Elmunzer BJ, Kim KJ, Lennon AM, Khashab MA, Kalloo AN, Singh VK. Incidence, severity, and mortality of post-ERCP pancreatitis: a systematic review by using randomized, controlled trials. Gastrointest Endosc. 2015 Jan;81(1):143-149.e9. doi: 10.1016/j.gie.2014.06.045. Epub 2014 Aug 1. PMID 25088919
- [Result] Kwak N, Yeoun D, Arroyo-Mercado F, Mubarak G, Cheung D, Vignesh S. Outcomes and risk factors for ERCP-related complications in a predominantly black urban population. BMJ Open Gastroenterol. 2020 Sep;7(1):e000462. doi: 10.1136/bmjgast-2020-000462. PMID 32943462
- [Result] Fujita K, Yazumi S, Matsumoto H, Asada M, Nebiki H, Matsumoto K, Maruo T, Takenaka M, Tomoda T, Onoyama T, Kurita A, Ueki T, Katayama T, Kawamura T, Kawamoto H; Bilio-pancreatic Study Group of West Japan. Multicenter prospective cohort study of adverse events associated with biliary endoscopic retrograde cholangiopancreatography: Incidence of adverse events and preventive measures for post-endoscopic retrograde cholangiopancreatography pancreatitis. Dig Endosc. 2022 Sep;34(6):1198-1204. doi: 10.1111/den.14225. Epub 2022 Feb 4. PMID 34963021
- [Result] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521